CLINICAL TRIAL: NCT06559449
Title: Cholecystectomy for Acute Cholecystitis During Weekend Compared to Delayed Weekday Surgery- a Nationwide Population Cohort Study
Brief Title: Cholecystectomy During Weekends
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: 10105555
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Acute Cholecystitis
Keywords: Cholecystitis; Emergency surgery; Laparoscopic cholecystectomy; Weekend surgery
MeSH Terms: conditions — Cholecystitis, Acute; Cholecystitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Weekend surgery: Patients undergoing surgery during weekend or national holiday
- Weekday group: Patients waiting in hospital during weekend and undergoing surgery during a weekday

SUMMARY:
Acute cholecystitis is the most common acute complication of gallstone disease. Although there are diverging opinions about optimal timing for surgery, the general recommendation is that surgery is performed as soon as possible after admission when the diagnosis is established. The study will compare acute cholecystectomies for acute cholecystitis performed during weekends with procedures where patient have been waiting during weekend and surgery performed during a subsequent weekday.

Hypothesis: Performing acute cholecystectomies for acute cholecystitis during weekends are associated with higher risk for complications.

DETAILED DESCRIPTION:
Acute cholecystitis is the most common acute complication of gallstone disease. About 15-20% of all cholecystectomies is performed because of acute cholecystitis. Laparoscopic cholecystectomy is one of the most common acute surgical procedure, and several studies have tried to identify the optimal time between debut of symptoms and surgery.

Although there are diverging opinions about optimal timing for surgery, the general recommendation is that surgery is performed as soon as possible after admission when the diagnosis is established. According to the latest Tokyo Guidelines, early laparoscopic cholecystectomy is the recommended treatment for all severity grades of acute cholecystitis, and delayed surgery is only recommended for selected high-risk patients. An English study based on data from a national register have shown that surgery within three days after admission is recommended for patients with acute cholecystitis. A randomised controlled trail (RCT) with the same formulation of question would need a large number of patients to reach sufficient power, which makes it impossible to perform a study of that kind during a reasonable time. An alternative to RCT studies is studies based on national register data which provides a large number of patients to achieve sufficient statistical power.

In daily clinical practice, there are often other acute surgical procedures with higher priority, leading to down prioritizing of acute cholecystectomies causing the surgery to be delayed. This is common despite that early cholecystectomy generally is accepted as golden standard for acute cholecystitis. Although there are sufficient evidence that risk for complication, days admitted at hospital and risk for conversion to open surgery are increased for every day that surgery is postponed, the phenomenon of delay is usual. To avoid delay of surgery, many clinics perform cholecystectomies during weekends and out-of-hours. Results from studies that compare complication rate between cholecystectomies performed during out-of-hours and office-hours are contradictive. This difference seems to be even larger for cholecystectomies that are performed during weekends, when there are often surgeons during internship and surgeons not specialized in upper GI-surgery on call. To this day, there are no published studies that investigates acute cholecystectomies following acute cholecystitis performed during weekend compared to operations that are delayed until the next following weekday.

The study will be a population-based cohort studie. Data will be extracted from the Swedish gallstone surgery and Retrograde Cholangiopancreatography register (GallRiks). The register is established and have collected data about patients undergoing cholecystectomies and ERCPs since 2005. More than 90% of all cholecystectomies and endoscopic retrograde cholangiopancreaticographies (ERCPs) performed in Sweden are registered. About 20 000 procedures (12 000 cholecystectomies and 8000 ERCPs) are annually registered, and data about indication for surgery, surgical technique, duration of surgery and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of ongoing acute cholecystitis.
* Undergoing surgery on a weekend or national holiday.
* Staying in hospital during weekend and undergoing surgery on any subsequent weekday.

Exclusion Criteria:

* Paediatric patients (<18 years)
* Patients who underwent surgery more than 7 days after admission
* Patients admitted and operated on during weekdays during the same week
* Patients with missing data regarding age, sex, American Society of Anesthesiologists Classification system (ASA grade), surgical approach, operating time, or complications.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cholecystectomy with ongoing acute cholecystitis that are registered in GallRiks (the Swedish Gallstone Surgery and ERCP register)
Sampling Method: Non-Probability Sample
Enrollment: 15730 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Complication rate | 30 days
  Number of patients with registered complications after surgery

SECONDARY OUTCOMES:
Open surgery | 30 days
  Number of surgical procedures completed with open technique (open or laparoscopic converted to open)
Prolonged surgery | 30 days
  Number of surgical procedures with operating time more than 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Umeå, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No